CLINICAL TRIAL: NCT00424112
Title: Stages an Processes of Change in Help-Seeking and Drinking Behavior
Brief Title: Motivation in Alcohol Treatment Facilities
Status: Completed | Type: Observational
Sponsor: University Medicine Greifswald (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Other Study IDs: E2_P1; 01EB0420
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Last update posted 2007-01-18 (Estimated); Status verified 2007-01

CONDITIONS: Alcohol Dependence; Alcohol Abuse
Keywords: motivation to change; treatment motivation; alcohol use disorders
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of this study is to determine if and to what extend a composite measure of treatment motivation and behavior change motivation predicts alcohol treatment success. It is expected that the composite measure based on the stages of the Transtheoretical Model of Behavior Change is a better predictor for treatment outcome than treatment motivation or behavior change motivation alone. Participants will be recruited from alcohol treatment centers. A baseline interview regarding their motivation, drinking behavior and personal treatment goals will be conducted. At the end of treatment, treatment staff will be asked about treatment involvement of each participant. Two follow-up interviews will be conducted after 6 and 12 months. To identify the impact of behavior change and treatment motivation on change in drinking behavior, data will be pooled with a non-treatment seeking sample. Conclusions can be drawn on what motivation pattern best predicts behavior change for those utilizing formal help and for those remitting without formal help (self-changers).

ELIGIBILITY:
Inclusion Criteria:

* Alcohol dependence
* Alcohol abuse

Exclusion Criteria:

* Persons physically and mentally not capable of participating in study

Ages: 18 Years to 64 Years | Sex: All
Age Groups: Adult
Enrollment: 450
Dates: Start 2004-10; Study Completion 2006-09

CONTACTS AND LOCATIONS:
Overall Officials: Jennis Freyer-Adam, Dr, Principal Investigator — University Medicine Greifswald; Ulfert Hapke, Dr, Principal Investigator — University of Applied Sciences Muenster; Ulrich John, Prof Dr, Study Director — University Medicine Greifswald
Locations (2):
- Germany (2):
  - Johnanna-Odebrecht-Stiftung, Greifswald, Mecklenburg-Vorpommern
  - Krankenhaus West, Stralsund, Mecklenburg-Vorpommern